CLINICAL TRIAL: NCT01526252
Title: Establishing a Reference Population for Normal Left Ventricular Function Parameters to Validate the Use of Two Dimensional Speckle Tracking Imaging Software in the Scar Study
Brief Title: Reference Population for Speckle Tracking Imaging
Acronym: STE Normal
Status: Completed | Type: Observational
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Terrence Ruddy, Principal Investigator, Ottawa Heart Institute Research Corporation
Other Study IDs: #2011803-01H
Record Dates: First submitted 2012-01-31; First posted 2012-02-03 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Left Ventricular Function
Keywords: speckle tracking echocardiography; database

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The SCAR study uses a software program entitled QLAB, a proprietory program, developed by Philips Healthcare (Philips Healthcare, Andover, MA). Literature on two-dimensional speckle tracking imaging (2DSTE) is growing, but data relevant to the population in the SCAR study is minimal. Accumulation of data relevant for a population of subjects will provide a set of normal values for interpretation of 2DSTE and minimize any influences from differences in data produced from different companies. This data may also assist other researchers investigate other cardiac diseases and abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 20 - 80 years at study entry
* Provide written informed consent and be able to comply with study procedures, including permission to access medical records
* Have a BMI index equal to or less than 35
* Less than 5% risk of developing coronary artery disease as determined using the Combined Diamond/Forrester and CASS data (ACC Stable CAD Guidelines)

Exclusion Criteria:

* Have taken cardioactive drugs within 6 months prior to examination

  * These include but are not limited to beta-blockers, calcium channel blockers, and angiotensin converting enzyme inhibitors
* Currently clinically significant chronic or acute illness
* Documented cardiovascular disease
* Possess abnormal cardiac structure and function after examination with routine ECHO

  * This may include valvular defects, left ventricular hypertrophy, cardiomyopathies or pericardial disease
* Documented congenital heart conditions or defects
* History of diabetes
* Be unwilling to provide voluntary consent

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal healthy males and females
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Establishment of normal values data in males and females aged 20 - 80 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Terrence Ruddy, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The objective of the trial was to establish a normal database for comparison. The database has not produced a specific study result. There is no publication as the sample size was not adequate.